CLINICAL TRIAL: NCT03214172
Title: Characterizing Recurrent Thromboembolism, Major Bleeding and All-Cause Death in Patients With Cancer-Associated Thromboembolism Treated With Rivaroxaban
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 19622
Record Dates: First submitted 2017-07-09; First posted 2017-07-11 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer-associated thrombosis: Adult patients with active cancer with at least one index venous thromboembolism (VTE) and no anticoagulation use during the 6-months (baseline period) prior to the index VTE event
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 15/20 mg

SUMMARY:
To estimate the real-world rates of recurrent Venous thromboembolism (VTE), major bleeding and all-cause mortality in patients with Cancer-associated thrombosis (CAT) treated with rivaroxaban

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years-of-age) with active cancer
* Patient with at least one index venous thromboembolism (VTE )
* ≥6-months of continuous eligibility prior to the index VTE event (baseline period).
* Newly initiated on rivaroxaban

Exclusion Criteria:

* Patients with any medical claim for Deep vein thrombosis (DVT) or Pulmonary embolism (PE) during the 6 months pre-index date
* Patients with prescription claim for anticoagulation therapy during the 6-month pre-index VTE period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Truven Health MarketScan Commercial Claims and Medicare Supplemental Databases is used. The Truven Health MarketScan® Research Databases capture person-specific clinical utilization, expenditures, and enrollment across inpatient, outpatient, prescription drug, and carve-out services. Individuals enrolled in the MarketScan databases are largely representative of the United States population in terms of age, sex, and type of health insurance coverage. The data come from a selection of large employers, health plans, and government and public organizations and contain claims from approximately 100 employers, health plans, and government and public organizations representing about 50 million covered lives across all age groups. The data elements to be used in the proposed study will include health plan enrollment records, participant demographics, inpatient and outpatient medical claims and outpatient prescription drug dispensing records.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Recurrent Venous thromboembolism | Retrospective analysis from November 2012 through September 2015
  Derived using inpatient and outpatient medical claims
Bleeding (based on the Cunningham algorithm) | Retrospective analysis from November 2012 through September 2015
  Derived using inpatient and outpatient medical claims
Mortality (In-hospital mortality or need for hospice care without subsequent healthcare claims) | Retrospective analysis from November 2012 through September 2015
  Derived using inpatient and outpatient medical claims

CONTACTS AND LOCATIONS:
Locations (1):
- US database, New York, New York, United States